CLINICAL TRIAL: NCT07028242
Title: Ultrasound and Histological Features of Patients With Atypical Endometrial Hyperplasia and Early Endometrioid Endometrial Carcinoma Submitted to Fertility Sparing Treatment.
Brief Title: Ultrasound and Histology in AEH and Early EEC Treated Conservatively
Acronym: ULTRA-SAFE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7691
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Fertility-Sparing Treatment (FST); Atypical Endometrial Hyperplasia; Early Endometrial Cancer (EEC)
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Intrauterine Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: This group includes patients with a histological diagnosis of atypical endometrial hyperplasia (AEH) or endometrioid endometrial carcinoma (EEC) G1-G2 who underwent hysteroscopic fertility-sparing surgery and medical treatment starting from January 2023. These patients were retrospectively identified from the Hysteroscopic Treatments Database. Only those with pre-treatment transvaginal ultrasound imaging available were included.
  Interventions: Procedure: Hysteroscopic fertility-sparing surgery and hormonal treatment
- Prospective: This group includes reproductive-age women newly diagnosed with AEH or EEC G1-G2, confirmed by endometrial biopsy during diagnostic hysteroscopy, who are eligible and consenting for fertility-sparing treatment. Patients undergo baseline clinical assessment, transvaginal ultrasound, and MRI prior to hysteroscopic surgery. Fertility-sparing treatment includes hysteroscopic endometrial resection, intrauterine device (IUD) placement and/or oral progestin therapy, followed by monitoring with serial biopsies and ultrasound at 3, 6, and 12 months.
  Interventions: Procedure: Hysteroscopic fertility-sparing surgery and hormonal treatment

INTERVENTIONS:
Procedure: Hysteroscopic fertility-sparing surgery and hormonal treatment — Patients undergo hysteroscopic endometrial resection using the Mazzon "three-step" technique or tissue removal device (TRD), depending on the lesion type. Following surgery, hormonal treatment is administered either via intrauterine device (IUD) or oral progestin. Monitoring includes serial endometrial biopsies and transvaginal ultrasounds at 3, 6, and 12 months.
  Other Names: Endometrial resection Hormonal therapy Intrauterine device (IUD) placement Oral progestin therapy

SUMMARY:
Ultra-S.A.F.E. is a multicenter, ambispective observational study investigating the ultrasound and histological characteristics of patients with atypical endometrial hyperplasia (AEH) or endometrioid endometrial carcinoma (EEC) G1-2 undergoing fertility-sparing treatment (FST). The study aims to describe pre-treatment ultrasound features, evaluate endometrial modifications during treatment, and assess histological and reproductive outcomes. It includes a prospective cohort (new patients recruited at three gynecologic oncology centers) and a retrospective cohort (patients treated conservatively since January 2023). Approximately 50 patients will be enrolled over 24 months, with clinical, ultrasound, and histological data collected. The ultimate goal is to enhance the diagnostic and monitoring role of transvaginal ultrasound (TVUS) in conservative treatment for fertility preservation.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18-45 years.

Histologically confirmed atypical endometrial hyperplasia (AEH) or endometrioid endometrial carcinoma (EEC) G1-2.

Candidates for fertility-sparing treatment (hysteroscopic resection and/or progestin therapy).

No prior history of invasive endometrial carcinoma.

Adequate endometrial visualization via transvaginal ultrasound (TVUS) and/or MRI.

Signed informed consent for study participation.

Exclusion Criteria:

Women under 18 or over 45 years.

Presence of myometrial invasion on MRI or histological analysis.

Histological diagnosis of serous carcinoma, clear cell carcinoma, or undifferentiated carcinoma.

History of previous hysterectomy or non-conservative surgical treatment.

Contraindications to hormonal therapy (e.g., thromboembolic disease, hormone-dependent malignancies).

Pregnancy at the time of enrollment.

Lack of adequate imaging for ultrasound-based assessment.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — The study is limited to female participants, as it investigates conditions affecting the endometrium. Eligibility is determined based on biological sex, rather than gender identity, due to the nature of the pathology and the focus on fertility-sparing treatment in patients with atypical endometrial hyperplasia (AEH) or endometrioid endometrial carcinoma (EEC) G1-2.
Study Population: The study population consists of women of reproductive age (18-45 years) diagnosed with atypical endometrial hyperplasia (AEH) or endometrioid endometrial carcinoma (EEC) G1-2, who are eligible for fertility-sparing treatment. Participants are recruited from three gynecologic oncology centers (Rome, Naples, and Turin) and classified into prospective (newly enrolled) and retrospective (previously treated since January 2023) cohorts.
  The study focuses on analyzing endometrial ultrasound features, assessing response to conservative therapy, and evaluating reproductive outcomes in patients undergoing hysteroscopic resection and/or progestin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-11 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Transvaginal ultrasound evaluation of the endometrium in patients with AEH or EEC G1-2 before fertility-sparing treatment | Baseline (pre-treatment), before hysteroscopic surgery and initiation of medical therapy.
  Analysis of pre-treatment ultrasound features of the endometrium and/or endometrial lesions, correlating findings with histological data and treatment outcomes.

SECONDARY OUTCOMES:
Endometrial ultrasound changes during medical treatment | Baseline, 6 months, and 12 months post-treatment initiation.
  Evaluation of ultrasound modifications of the endometrium throughout conservative treatment, correlated with hysteroscopic and histological findings.
Ultrasound predictors of treatment response | Baseline and 6 months post-treatment.
  Comparison of pre-treatment ultrasound features between patients who achieve remission and those with persistent disease after 6 months of therapy.
Endometrial ultrasound characteristics and reproductive success | Baseline and 12 months post-treatment
  Analysis of pre-treatment ultrasound features in patients who achieve pregnancy versus those with negative reproductive outcomes within 12 months of treatment
Correlation between ultrasound and molecular profiling | Baseline
  Investigation of potential associations between endometrial ultrasound characteristics and molecular markers of atypical endometrial hyperplasia or endometrial carcinoma
Comparison of ultrasound and MRI findings | Baseline
  Assessment of ultrasound imaging in comparison to MRI for pre-treatment evaluation of endometrial lesions

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Carla Testa, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy